CLINICAL TRIAL: NCT04807686
Title: Attenuation of Tonal Tinnitus by Lateral Inhibition Therapy
Acronym: TIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Dr Quemar (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018-A02448-47
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional algorithm (Active Comparator)
  Interventions: Device: Auditory simulation
- notched-type algorithm (Experimental)
  Interventions: Device: Auditory simulation

INTERVENTIONS:
Device: Auditory simulation — Each patient will be delivered each of the 2 auditory stimulation protocols considered in the context of the research: stimulation with a traditional algorithm called AT and stimulation with a notched-type algorithm called AE. The order in which will be carried out, for the same patient, each of these 2 protocols (AT then AE or AE then AT) will be randomized.

SUMMARY:
Lateral Inhibition Therapy (TIL) corrects the patient's hearing by notched amplification on the patient's listening soundtrack. This half-octave notch is targeted at tinnitus frequencies measured tonal. The device slightly increases the amplification around the notch, so that the cerebral cortex compensates for this "gap" in the sound spectrum, masking the crippling tinnitus at the same time. This research is based on a new algorithm developed by the SIEMENS Company which proposes an attenuation of tonal tinnitus by a TIL by notched amplification emitted by the hearing device, object of the study.

DETAILED DESCRIPTION:
In France, up to 16 million people suffer from tinnitus or ringing in the ears daily. This parasitic sound that does not come from the patient's environment can interfere with each individual in a variable way, sometimes creating an insurmountable handicap which has not known any effective treatment validated to date.

Lateral Inhibition Therapy (TIL) corrects the patient's hearing by notched amplification on the patient's listening soundtrack. This half-octave notch is targeted at tinnitus frequencies measured tonal. The device slightly increases the amplification around the notch, so that the cerebral cortex compensates for this "gap" in the sound spectrum, masking the crippling tinnitus at the same time. This research is based on a new algorithm developed by the SIEMENS Company which proposes an attenuation of tonal tinnitus by a TIL by notched amplification emitted by the hearing device, object of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old.
* Patient with disabling tonal tinnitus (THI score> 40) for more than 6 months.
* Patient with a hearing loss of at least 25dB, centered on the frequency of tinnitus and requiring hearing aids
* Patient who has never used a hearing aid or a tinnitus masking system.
* Patient who stopped all tinnitus treatment at least 1 month before the start of the study (drug treatment, psychotherapy).
* Patient being willing to attend all of the visits planned as part of the study.
* Patient affiliated or beneficiary of a social security scheme.
* Patient having signed the free and informed consent

Exclusion Criteria:

* Minor patient.
* Patient with hyperacusis
* Patient already with a hearing aid or tinnitus masker.
* Patient undergoing psychotropic or neurotropic drug treatments.
* Patient with a history of psychological or psychiatric disorders.
* Patient with a contraindication to wearing hearing aids.
* Patient suffering from non-disabling tinnitus (THI score <40).
* Patient suffering from intermittent, non-tonal or pulsatile tinnitus.
* Patient participating in another clinical study.
* Protected patients: adults under guardianship, curatorship or other legal protection, deprived of their liberty by judicial or administrative decision.
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2019-07-19 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory | 2 months
  The primary endpoint is the score (out of 100 points) obtained on the Tinnitus Handicap Inventory (THI), expressed in terms of variation from the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Quemar, Doctor, Principal Investigator — Ramsay santé
Locations (1):
- Hôpital Privé Clairval, Marseille, France